CLINICAL TRIAL: NCT00370500
Title: Quetiapine and the Dopaminergic Epigenetic Control - a Pilot Study
Brief Title: Quetiapine and the Dopaminergic Epigenetic Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Stefan Bleich, University of Erlangen-Nürnberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D1449L00029; EudraCT-Nr: 2005-006151-20
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Dopamine transporter gene; DNA methylation; Epigenetics
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): There is only one arm in this study. All probands receive quetiapine.
  Interventions: Drug: Quetiapine fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate — Dosage and frequency are judged by the study physician. The dosage must not excess 800mg/d.
  Other Names: Seroquel(R)

SUMMARY:
BACKGROUND:

Epigenetic modifications such as DNA-methylation and histone acetylation are known to be involved in the pathophysiology of schizophrenia. Aim of the present study is to investigate

1. whether differences in the methylation pattern of the promoters of dopaminergic genes exist between schizophrenic patients and healthy controls and
2. whether treatment with the second generation antipsychotic quetiapine leads to changes in the methylation pattern of those genes in patients suffering from schizophrenia.

STUDY DESIGN AND METHODS:

50 male patients and 50 male controls are to be enrolled into the study. Patients will be treated with quetiapine for 3 weeks. Blood samples will be drawn before treatment and after three weeks to measure DNA-methylation status. Clinical characterisation includes PANSS, AIMS, BDI. Healthy probands will not be treated.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study subjects must fulfil all of the following criteria:

1. Provision of written informed consent
2. A diagnosis of schizophrenia by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
3. Able to understand and comply with the requirements of the study
4. Age 18 - 65 years

Exclusion criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Any DSM-IV Axis I disorder not defined in the inclusion criteria
2. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
3. Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
4. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
5. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
6. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before inclusion
7. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
8. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
9. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
10. Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
11. Involvement in the planning and conduct of the study
12. Previous enrolment in the present study.
13. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
14. Actual treatment with clozapine or clozapine treatment during the previous three month. Other antipsychotic drugs will be allowed, if intake can be terminated during the two day wash out period.
15. Previous history of major head injuries or neurological disorders
16. Intake of homocysteine lowering vitamins (folate, B12, B6)
17. Renal failure
18. Intake of nutritional derivatives which influence epigenetic patterns (butyrate from milk products, tea polyphenol or epigallo-catechin-3-gallate which inhibits DNMT)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Primary variable is the amount of methylated vs. unmethylated promoter specific DNA in the DAT gene of patients before and after treatment with quetiapine (within group comparison). | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bleich, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Department of Psychiatry and Psychotherapy, University Erlangen-Nuremberg, Erlangen, Germany